CLINICAL TRIAL: NCT05847972
Title: Evaluation of the Effect of Manual Therapy and the Application of Plantar Orthoses in Amateur Runners With Ankle Range of Motion Restriction. A Randomised Clinical Trial.
Brief Title: Effect of Manual Therapy and Inmediately Application of Plantar Orthoses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCV/2022-2023/093
Record Dates: First submitted 2023-04-05; First posted 2023-05-08 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Ankle Injuries and Disorders
Keywords: ankle; plantar orthoses
MeSH Terms: conditions — Ankle Injuries; Disease | interventions — Movement

STUDY DESIGN:
Who Masked: Participant
Masking Description: The groups will be arranged randomly and the masking technique to be used will the single blind procedure. The random allocation to each group will be made just by the software Epidat version 4.2 of the Galician Health Service (link: https://www.sergas.es/Saude-publica/EPIDAT?idioma=es).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): A will undergo MWM and have their moulds taken in phenolic foam immediately after the musculoskeletal manipulation.
  Interventions: Procedure: MWM (Mobilization with movement); Device: Plantar orthoses
- Control Group (Placebo Comparator): Participants will undergo MWM and moulds will be taken one week after the musculoskeletal manipulation.
  Interventions: Procedure: MWM (Mobilization with movement); Device: Plantar orthoses

INTERVENTIONS:
Procedure: MWM (Mobilization with movement) — This manipulation is intended to improve ankle dorsiflexion. One session of 3 sets of 20 slow ankle dorsiflexion's separated by 10 seconds of rest will be performed.
Device: Plantar orthoses — Procedure: MWM All participants will undergo MWM. This manipulation is intended to improve ankle dorsiflexion. One session of 3 sets of 20 slow ankle dorsiflexion's separated by 10 seconds of rest will be performed.
  Procedure: Plantar orthoses The moulds will be taken immediately after the manipulation. The PO will be made of resin (0.8mm +1.2mm), 2mm hard EVA heel stabiliser, 3mm semi-hard EVA cover. The PO should be worn for 3 months to obtain the results of the study.

SUMMARY:
Limitation of ankle dorsiflexion is directly related to pronated foot. For its treatment, plantar orthoses and manual therapy are used. There is a lack of evidence on their combination, as to when the cast should be taken after manipulation. Our hypothesis proposes that it is more effective to cast immediately after manipulation.

DETAILED DESCRIPTION:
The popularity of long-distance running has increased because it can be practised in many settings, the low cost and the links to prevention of health problems. In running between 19-79% of runners may suffer a running-related overuse injury each year. Pronated feet have been identified as a risk factor for lower limb overuse injury, and several studies have found that ankle dorsiflexion limitation is related to pronated feet.

There is a lack of evidence on their combination, as to when the cast should be taken after manipulation. Our hypothesis proposes that it is more effective to cast immediately after manipulation.

The main objective is to compare the effect of manipulation with motion (MWM) performed immediately prior to casting for plantar orthoses (PO) with the effect of manipulation with motion performed one week prior to casting for plantar orthoses on ankle dorsiflexion (ankle DF) and foot pronation in runners with hyper pronator feet secondary to a limited ankle DF.

This study's population will be composed by at least 16 individuals per group, both male and female, with ages among 18 and 45.

They will be randomised into two groups; group A, which will undergo MWM and have the moulds taken in phenolic foam immediately after the manipulation. The other group will be group B, which will undergo the MWM, and the moulds will be taken one week after the manipulation.

ELIGIBILITY:
Inclusion Criteria:

* Runners who run on asphalt.
* Individuals who run at least >6 hours per week for 6 months prior to study participation.
* Participants with hyperpronated feet secondary to ankle ROM limitation.
* Runners with an ankle DF difference of >1.5cm in both feet or an ankle DF of less than 11.5cm according to the Lunge Test.

Exclusion Criteria:

* Individuals who have suffered a major injury in the previous two months.
* FPI less than 6.
* Runners wearing minimalist footwear into which PO cannot be inserted.
* Individuals already undergoing treatment with plantar supports.
* Chronic widespread pain, including fibromyalgia.
* Systemic rheumatic pathologies.
* History of recent trauma or surgery

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline dynamic degrees of ankle dorsiflexion at 12 weeks | At baseline; post 1 (inmmediate); post 2 (3weeks); post 3 (6weeks) and post 4 (12weeks)
  Measured with Kinovea software. The patient will be recorded running in slow motion and the peroneal malleolus, the centre of the heel by the lateral edge and the head of the V metatarsal will be marked. It will then be analysed using Kinovea software

SECONDARY OUTCOMES:
Degrees of DF of the ankle in closed kinetic chain with the Lunge Test using LegMotion | At baseline; post 1 (inmmediate); post 2 (3weeks); post 3 (6weeks) and post 4 (12weeks)
  Lung Test will measure the distance between the toes and the Legmotion stirrup, which has been shown to have a moderate to excellent intra-rater reliability (ICC = 0.65-0.99) with a minimum detectable change of 1.9 cm and 4.7°.
Degrees of pronation in dynamics, measured with Runscribe (DP) | At baseline; post 1 (inmmediate); post 2 (3weeks); post 3 (6weeks) and post 4 (12weeks)
  Runsribe sensors will be placed on the runners while they run. Data will be recorded with the official Runscribe App. This method is validated by Lewin et al.
Foot Function Index | At baseline; post 1 (inmmediate); post 2 (3weeks); post 3 (6weeks) and post 4 (12weeks)
  FFI for the assessment of pain, disability and limitation of foot function, recommended for use in both clinical and research settings.

CONTACTS AND LOCATIONS:
Locations (1):
- Juan Vicente-Mampel, Torrent, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No